CLINICAL TRIAL: NCT04563208
Title: A Randomized, Double-Blind, Study Comparing the Efficacy, Safety, and Tolerability of Oral Administration of Ribavirin (RBV) and Nitazoxamide (NTZ)Versus Placebo in SARS-CoV-2 Virus Infected Participants (DuACT)
Brief Title: Study of Oral Administration of Ribavirin and Nitazoxamide Versus Placebo in COVID-19
Acronym: DuACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Collaborators: SynaVir (Industry)
Responsible Party: Principal Investigator, Professor Francois Venter, Divisional Director: Ezintsha, University of Witwatersrand, South Africa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DUACT-101
Record Dates: First submitted 2020-09-21; First posted 2020-09-24 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Covid19; SARS-CoV Infection
Keywords: Ribavirin; Nitazoxanide; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Placebo (Placebo Comparator): Placebo administered
  Interventions: Drug: Placebo
- Arm B: Ribavirin/Nitazoxanide (RBV/NTZ) (Active Comparator): Ribavirin/Nitazoxanide (RBV/NTZ) administered
  Interventions: Drug: DuACT

INTERVENTIONS:
Drug: Placebo — Placebo administered on Days 1-5
  Arms: Arm A: Placebo
Drug: DuACT — Day1: RBV 600 mg BID and NTZ 500 mg BID Days 2-5: RBV 400 mg BID and NTZ 500 mg BID
  Arms: Arm B: Ribavirin/Nitazoxanide (RBV/NTZ)

SUMMARY:
This is a single center, randomized, double-blind, 2-arm, parallel-group study of DuACT in participants with clinical symptoms of COVID-19 that have begun within the past 72 hours prior to testing.

DETAILED DESCRIPTION:
This is a single center, randomized, double-blind, 2-arm, parallel-group study of DuACT in participants with clinical symptoms of COVID-19 that have begun within the past 72 hours prior to testing. A confirmatory diagnosis of COVID-19 via nasopharyngeal swab, with a positive PCR result within 48 hours of testing.

Consented participants who complete screening and meet study eligibility criteria will be randomized in a 1:1 ratio to receive DuACT or Placebo for 5 days.

Study drugs will be administered BID for 5 days with a loading dose on Day 1. Following randomization, participants will complete a symptom questionnaire, record temperature and record oxygen saturation daily for 10 days and at day 28. A thermometer and pulse oximeter will be provided to each patient at the baseline visit (Day 1).

On study days 3, 6 and 10 participants will have a clinic or home visit by a home healthcare provider. At these visits, a mid-turbinate nasal swab will be obtained, confirmation of the patient's clinical symptoms questionnaire will be completed and any adverse events will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Signed a current EC approved informed consent form
2. Male or female participants between 18 and 75 years of age, inclusive diagnosis of SARS-CoV-2 infection, with all of the following, with onset of any within the 72 hours prior to testing:

   1. Presence of fever at time of screening of ≥ 38.0°C (≥ 100.0°F) and/or
   2. Presence of at least one constitutional symptom associated with Covid-19 (e.g. headache, myalgia, malaise, or fatigue, rash, diarrhea, loss or alteration of taste/smell) of any severity, and/or
   3. Presence of at least one respiratory symptom (e.g. cough, chest tightness or sore throat) and/or
3. Diagnosis of COVID-19 with a positive PCR in the past 48 hours

Exclusion Criteria:

1. Pregnant or lactating females
2. Critically ill with presence of one or more of the following signs:

   1. difficulty breathing or shortness of breath
   2. need for admission to a hospital or an intensive care unit,
   3. acute respiratory failure requiring intubation/mechanical ventilation,
   4. signs of shock including hypotension
   5. Oxygen saturation < 92 %
3. Any clinically significant screening laboratory results that are greater than 5 times the upper limit of normal.
4. Estimated GFR < 50 mL/min/1.73 m2 (calculated using either Modification of Diet in Renal Disease (MDRD) or Cockcroft Gualt
5. Known genetic hemoglobinopathy (e.g., thalassemia major or sickle cell anemia) or autoimmune hemolytic anemia
6. Hemoglobin less than 10 gm/dL or hematocrit < 30 %
7. Retinal eye disease
8. Known chronic kidney disease, stage - 5 or receiving dialysis
9. Inability to tolerate oral medications
10. Allergy or prior adverse reaction to either ribavirin or nitazoxanide
11. QTc interval > 450 mSEC for men and women
12. History of Torsade de Pointes VT or prior cardiac arrest or congenital long QT interval
13. Current treatment with histamine-2 receptor antagonists (H2 blockers) and/or Protein Pump Inhibitors and throughout the study.
14. Have been vaccinated against COVID-19
15. Have participated in a clinical study in the past 30 days
16. Any physical, mental, or social condition, drug/alcohol use, history of illness or laboratory abnormality that in the investigator's judgment might interfere with study procedures or the ability of the subject to adhere to and complete the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Rate of decline in viral load | 10 days
  Rate of decline in viral load over the 10 days after randomization between participants treated with RBV and NTZ for COVID-19 and placebo

SECONDARY OUTCOMES:
Time to resolution of viral load | 28 days
  Time to resolution of viral load, defined by reduction of virus below LLOQ and maintaining it for 2 days.
Comparison of proportion of subjects who are asymptomatic and symptomatic | 10 days
  Comparison of proportion of subjects who are asymptomatic and symptomatic at day 10
Rate of decline in viral load | Days 3 and 6
  To assess the rate of decline in viral load over days 3 and 6 after randomization
Change in modified NEWS-2 | 28 days
  Assess change in modified National Early Warning System-2 items on a scale of 0 to 20. HIgher scores meaning greater clinical risk.
Proportion of subjects with treatment emergent adverse events | 28 days
  Proportion of subjects with treatment emergent adverse events leading to study drug discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Simiso Sokhela, Principal Investigator — Ezintsha
Locations (1):
- Sunnyside Office Park, Johannesburg, Gauteng, South Africa